CLINICAL TRIAL: NCT02006979
Title: The Effects of Exercise Before Doxorubicin Chemotherapy on Cardiac Function
Brief Title: Acute Exercise Cardioprotection From Doxorubicin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Kristin Campbell, Dr. Kristin Campbell, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H13-03090
Record Dates: First submitted 2013-12-05; First posted 2013-12-10 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Breast Cancer
Keywords: cardiotoxicity; Chemotherapy, Adjuvant; Breast Neoplasms; Exercise; Cardiotoxins; Echocardiography; Speckle tracking; Biological Markers; Electrocardiography
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): an acute bout of exercise performed ≤24 hours prior to each cycle of anthracyclines and no exercise for 48 hours post
  Interventions: Other: exercise
- No exercise (No Intervention): no exercise for 72 hours prior or 48 hours post each cycle of anthracyclines

INTERVENTIONS:
Other: exercise — An acute bout of exercise performed 24 hours prior to every anthracycline infusion.
  Arms: Exercise

SUMMARY:
In rodents, a single bout of exercise prior to injection of a chemotherapy agent used to treat breast cancer prevents or attenuates a number of markers of cardiac injury. This study will investigate whether this finding translates to human breast cancer patients. Participants scheduled to receive chemotherapy for breast cancer will be randomized to exercise or no exercise 24 hours prior to every chemotherapy treatment. The effect on cardiac function will be compared between groups noninvasively by echocardiography and electrocardiography and a venous blood draw at baseline before chemotherapy, after the first treatment and at the end of chemotherapy.

DETAILED DESCRIPTION:
1. Purpose The purpose of this study is to investigate whether performing a single bout of exercise 24 hours prior to receiving infusions of the anthracycline chemotherapy agent doxorubicin for breast cancer can prevent some of the damaging cardiac effects. Currently, doxorubicin is the most effective chemotherapy agent for breast cancer but is also the most damaging. As such, increased risk of cardiovascular disease is a growing concern in doxorubicin-treated patients. Current strategies for minimizing cardiac injury are dose reduction and discontinuation of therapy, which compromise the effectiveness of the treatment. Interventions that can minimize the cardiac injury associated with doxorubicin could reduce cancer-related and cardiovascular disease-related mortality in women diagnosed with breast cancer.
2. Hypotheses 1. Performing an acute bout of exercise within 24 hours before anthracycline infusion will decrease the acute negative change in subclinical markers of cardiotoxicity after the first anthracycline infusion seen in those who do not exercise for 72 hours prior.

2. Performing exercise within 24 hours before every infusion of anthracycline will decrease the negative change in markers of cardiac dysfunction seen at the end of chemotherapy in those who do not exercise for 72 hours prior to each infusion.

3) Justification An acute exercise bout prior to induction of a myocardial infarction in animals provides cardioprotective benefit by reducing the size of the infarct relative to control animals. Recently, acute exercise performed 24 hours before anthracycline injection in rodents has also provided a cardioprotective benefit. Oxidative stress and apoptosis of cardiomyocyte mitochondria are primary mechanisms of anthracycline-induced cardiotoxicity. The single acute bout of exercise prevented or attenuated some of the anthracycline-induced negative effects on cardiomyocytes including oxidative stress, apoptosis, mitochondrial dysfunction, as well as systolic dysfunction. There are no studies to date that have investigated the cardiac effects of an acute bout of exercise in close proximity to anthracycline infusion in humans. Aerobic exercise training is recommended throughout chemotherapy treatment, but there are no guidelines in place in terms of the timing of exercise in relation to receipt of chemotherapy infusions.

4) Objectives

1. To compare the acute effect of performing exercise (within 24 hours before the first infusion) compared to no exercise (no exercise for 72 hours prior to the first infusion) on markers of subclinical cardiotoxicity 24-48 hours after the first anthracycline infusion.
2. To compare the chronic effect of performing exercise (within 24 hours before every infusion) compared to no exercise (no exercise for 72 hours prior to every infusion) on markers of cardiotoxicity 7 to 14 days after the final anthracycline infusion 5) Research Method This study will be a two-arm randomized control trial. Twenty-four women aged 18 or older newly diagnosed with stage I-IIIA breast cancer, and scheduled to receive neoadjuvant or adjuvant doxorubicin chemotherapy in cycles of 2-3 weeks will be recruited by oncologist referral and posters. Participants will be randomized to one of two conditions: i) an acute bout of exercise performed ≤24 hours prior to each cycle of anthracyclines and no exercise for 48 hours post; or ii) no exercise for 72 hours prior or 48 hours post each cycle of anthracyclines.

6) Statistical Analysis The primary outcome will be global longitudinal strain measured by echocardiography. The secondary outcomes will be the NT-proBNP and cardiac troponin T cardiac biomarkers measured with an assay of blood taken via venous blood draw, echocardiography-derived left ventricular twist. The exploratory outcome measure will be treatment symptoms as reported by the Rotterdam Symptom Checklist. Cardiac outcome measures will be performed at the following time points: 1) Post diagnosis and prior to the first cycle of anthracyclines; 2) 24-48 hours after the first cycle; 3) at least one week after the last cycle of anthracyclines, but before subsequent chemotherapy treatments. The Rotterdam will be performed at baseline and within the last few days of each treatment cycle.

Baseline characteristics of the two groups will be compared with independent t-tests. Descriptive statistics and frequencies will be calculated for all continuous and categorical variables. The acute effect will be determined by the difference between time points 1) and 2). The chronic effect will be determined by the difference between time points 1) and 3). For each analysis, a linear mixed model with time as a fixed and repeated effect, group as a fixed effect, and a time by condition (2 x 2) interaction will be used. If the interaction effect is not statistically significant, the main effects of time and condition will be explored. An alpha of 0.05 will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed with stage I-IIIA breast cancer
* scheduled to receive neoadjuvant or adjuvant doxorubicin chemotherapy in cycles of 2-3 weeks long
* receive their oncologist's approval to exercise
* be able to complete first time point of data collection prior to first chemotherapy cycle
* be able to understand and provide written informed consent in English

Exclusion Criteria:

* concurrent participation in a structured exercise program or study
* have orthopedic limitations to exercise
* pre-existing cardiovascular disease
* uncontrolled hypertension (blood pressure ≥ 140/90 mmHg)
* uncontrolled diabetes
* respiratory disease
* current smoking status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin L Campbell, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Breast Cancer Research Exercise Gym, Vancouver, British Columbia, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: no exercise for 72 hours prior or 48 hours post each cycle of anthracyclines
Period: Overall Study
Arm/Group | Exercise | Usual Care
Started | 14 | 13
Completed | 13 | 11
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant in the usual care group did not complete baseline assessment. One participant in usual care group completed baseline assessment before protocol violation (did not receive any of study drug) and was excluded. One participant in the exercise group withdrew immediately after the baseline assessment and did not start the intervention.
Groups:
- Exercise: an acute bout of exercise performed ≤24 hours prior to each cycle of anthracyclines and no exercise for 48 hours post exercise
- Total: Total of all reporting groups
Arm/Group | Exercise | Usual Care | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (9) | 50 (10) | 50 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 7 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 13 | 11 | 24
Body weight [Mean (Standard Deviation); unit: kg] | 69.7 (11.7) | 72.2 (12.7) | 71.9 (12.7)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 13.0 (1.0) | 12.7 (1.1) | 12.8 (1.0)
6-month MVPA [Median (Full Range); unit: average weekly minutes] | 214 [0 to 701] | 124 [0 to 619] | 165 [0 to 701]
LVEF [Mean (Standard Deviation); unit: %] | 57 (4) | 58 (3) | 58 (3)
Cardiac output [Mean (Standard Deviation); unit: L/min] | 3.2 (0.6) | 3.0 (0.5) | 3.1 (0.5)
Resting HR [Mean (Standard Deviation); unit: beats per minute] | 69 (11) | 69 (12) | 69 (11)
Systemic vascular resistance [Mean (Standard Deviation); unit: dynes·sec·cm-5] | 1933 (445) | 2074 (514) | 1998 (472)
E/A ratio [Mean (Standard Deviation); unit: no units] | 1.20 (0.37) | 1.27 (0.32) | 1.23 (0.34)
Mean arterial pressure [Mean (Standard Deviation); unit: mmHg] | 75 (10) | 76 (11) | 76 (11)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 25.0 (4.8) | 26.7 (5.1) | 25.8 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Global Longitudinal Strain
Description: Assessed with 2D speckle tracking echocardiography
Time Frame: 24-48 hours after first doxorubicin and 7-14 days after completion of last doxorubicin cycle
Measure: Mean (Standard Deviation); unit: % deformation
Arm/Group | Exercise | Usual Care
Number analyzed (Participants) | 13 | 11
% deformation
  Baseline | 19.2 (1.9) | -19.6 (1.9)
  24-48 h post first doxorubicin | 21.4 (1.8) | -21.5 (1.6)
  7-14 days post last doxorubicin | -18.7 (1.4) | -20.3 (1.6)

2. Secondary Outcome: NT-proBNP
Description: biomarker of cardiac injury
Time Frame: 24-48 hours after first doxorubicin and 7-14 days after completion of last doxorubicin cycle
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Exercise | Usual Care
Number analyzed (Participants) | 13 | 11
pg/mL
  Baseline | 52 (30) | 59 (35)
  24-48 h post first doxorubicin | 214 (77) | 323 (151)
  7-14 days post last doxorubicin | 106 (78) | 77 (39)

3. Secondary Outcome: Cardiac Troponin T
Description: biomarker of cardiac injury
Time Frame: 24-48 hours after first doxorubicin and 7-14 days after completion of last doxorubicin cycle
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Exercise | Usual Care
Number analyzed (Participants) | 13 | 11
pg/mL
  Baseline | 1.3 (2.1) | 1.5 (2.3)
  24-48 h post first doxorubicin | 2.6 (3.2) | 1.9 (2.6)
  7-14 days post last doxorubicin | 13.6 (11.2) | 11.6 (8.3)

4. Secondary Outcome: LV Twist
Description: Assessed with 2D speckle tracking echocardiography
Time Frame: 24-48 hours after first doxorubicin and 7-14 days after completion of last doxorubicin cycle
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Exercise | Usual Care
Number analyzed (Participants) | 13 | 11
degrees
  Baseline | 16.4 (7.6) | 16.4 (5.9)
  24-48 h post first doxorubicin | 20.3 (8.5) | 22.4 (7.8)
  7-14 days post last doxorubicin | 15.7 (6.5) | 15.6 (6.6)

5. Other Pre Specified Outcome: Patient-reported Symptoms
Description: As assessed by standardized scores of physical and psychological distress by the Rotterdam Symptom Checklist
Time Frame: <1 week before the first doxorubicin, <3 days before the 2nd, 3rd, and 4th doxorubicin, 7-14 days after completion of the last doxorubicin cycle
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: During intervention period which lasted from shortly prior to the first doxorubicin treatment to 7-14 days after the last doxorubicin treatment.
Description: Serious adverse events related to the study intervention.
Arm/Group | Exercise | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No